CLINICAL TRIAL: NCT06693713
Title: The Youth Series Sanctuary Mental Health Ministries Randomized Control Trial
Brief Title: Sanctuary Youth Series Randomized Control Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanctuary Mental Health Ministries (Other)
Collaborators: Excellence in Giving Insights (Unknown)
Responsible Party: Principal Investigator, Kate Williams, Chief Impact Officer, Sanctuary Mental Health Ministries
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pending
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Mental Health; Mental Health Help-Seeking; Mental Health Literacy
Keywords: Mental Health; Youth
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilot Group (Experimental): This group will receive an 8 week course on mental health knowledge. The series has been designed as an eight-week program for youth ages 11-15 that uses games, short films, discussion questions, and exercises to engage with mental health and faith topics.
  Interventions: Other: Mental Health Youth Series
- Comparison Group (No Intervention): This group will not receive any mental health information, but will continue using their normal youth group material as planned. They will participate in the baseline and end line surveys.

INTERVENTIONS:
Other: Mental Health Youth Series — The Mental Health Youth Series is an eight-week program for youth ages 11-15 that uses games, short films, discussion questions, and exercises to engage with mental health and faith topics. The intervention package includes a facilitation guide and a guide for parents and caregivers. The program is intended to be conducted by an experienced facilitator, although there is no specific training provided for facilitators outside of the facilitation guide.
  Arms: Pilot Group

SUMMARY:
Sanctuary Mental Health Ministries designed an eight-week program for youth ages 11-15 that uses games, short films, discussion questions, and exercises to engage with mental health and faith topics. The intervention package includes a facilitation guide and a guide for parents and caregivers. The program is intended to be conducted by an experienced facilitator, although there is no specific training provided for facilitators outside of the facilitation guide. The facilitator would lead groups of 11-15 year olds by leading games, showing the films, and facilitating discussion. The series is freely available on Sanctuary's website; individuals can access the material by creating an account, logging in, and downloading the course content. This RCT is to evaluate the effectiveness of the Youth Series course on improving youth's mental health literacy, knowledge, and attitudes towards help-seeking.

DETAILED DESCRIPTION:
Churches will be recruited to the study based on social media sites and through Sanctuary's newsletter distribution lists. Churches who agree to participate in the study will be randomized to one of two groups, the Pilot Group that receives the 8-week series, and the Comparison Group, that does not receive the series. Both groups will be asked to complete a baseline survey and then a follow-up (end line) survey 8-weeks later. The results will be scored and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Youth between the ages of 11-18 attending a youth group that has been recruited to the study.

Exclusion Criteria:

* Youth outside of the age range that are not attending a youth group recruited to the study.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-11-18 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Mental Health Knowledge | 8 weeks
  Participants will answer mental health knowledge scores, either correct or incorrect.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Williams, Masters, Principal Investigator — Excellence in Giving Insights; Ashley Williams, Masters, Study Director — Excellence in Giving Insights; Lincoln Lau, PhD, Study Chair — University of Toronto
Locations (1):
- Excellence in Giving Insights, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to publish this data in the International Committee of Medical Journal (ICMJ)